CLINICAL TRIAL: NCT05396898
Title: Conversion to Extended-release MeltDose® Tacrolimus After Kidney Transplantation - Impact on Glucose Metabolism and Lipid Profile
Brief Title: Tacrolimus Formulation and Glucose Metabolism After Kidney Transplantation (TAGLUMET Trial)
Acronym: TAGLUMET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TAGLUMET
Record Dates: First submitted 2022-05-17; First posted 2022-05-31 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Posttransplant Diabetes Mellitus
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LCP-tacrolimus (Envarsus®) (Experimental): Patients in this arm start (after randomization) on LCP-tacrolimus therapy.
  At midterm of study participation (16 weeks), a switch is made to twice-daily tacrolimus (Prograf® ) therapy.
  The duration of the trial for each subject is expected to be 32 weeks.
  Interventions: Drug: LCP-tacrolimus
- twice-daily tacrolimus (Prograf®) (Active Comparator): Patients in this arm start (after randomization) on twice daily tacrolimus (Prograf®) therapy.
  At midterm of study participation (16 weeks), a switch is made to LCP-tacrolimus (Envarsus®) therapy. The duration of the trial for each subject is expected to be 32 weeks.
  Interventions: Drug: twice-daily tacrolimus

INTERVENTIONS:
Drug: LCP-tacrolimus — Prophylaxis of transplant rejection in liver and kidney allograft recipients
  Other Names: Envarsus®
  Arms: LCP-tacrolimus (Envarsus®)
Drug: twice-daily tacrolimus — Prophylaxis of transplant rejection in liver, kidney or heart allograft recipients
  Other Names: Prograf®
  Arms: twice-daily tacrolimus (Prograf®)

SUMMARY:
Posttransplantation diabetes mellitus after kidney transplantation mediated by tacrolimus is mainly dependent on dose and peak plasma concentration. To substantiate the potential benefits on glucose metabolism and lipid profile of LCP-tacrolimus compared to standard twice-daily tacrolimus after kidney transplantation, a prospective randomized intraindividual cross-over conversion trial with a comprehensive assessment of glucose metabolism and lipid profile is performed. Primary endpoint is the difference in insulin secretion between treatments, as the principal parameter affected by tacrolimus peak concentrations.

Aim of the study is, to assess glucose metabolism under different tacrolimus formulations (LCP-tacrolimus and twice-daily tacrolimus).

DETAILED DESCRIPTION:
Posttransplantation diabetes mellitus (PTDM) is an increasing problem in solid organ transplantation with profound impact on patient and allograft survival. One major contributing factor for the development of PTDM is choice of immunosuppression. Calcineurin inhibitors (CNIs), especially tacrolimus display a substantial diabetogenic potential but remain a cornerstone in maintenance immunosuppression for prevention of rejection and allograft loss. The diabetogenic effect of tacrolimus is mediated predominantly via disturbance of beta-cell function and impaired insulin secretion. There is growing evidence that this effect is dependent on dose and peak plasma concentrations. Once-dailyLCP-tacrolimus has been shown to have lower peak concentrations than twicedaily tacrolimus with comparable efficacy and safety.

LCP-tacrolimus has been shown to improve triglyceride levels, compared to twicedaily tacrolimus. In this study, no effect on the incidence of PTDM was observed, however assessed only by fasting plasma glucose, HbA1c and antidiabetic treatment. As 1/3 of patients with diabetes are solely diagnosed via oral glucose tolerance test, this approach is insufficient for proper evaluation of glucose metabolism, including prediabetes as the principal risk factor.

From pathophysiologic understanding blood lipids and glucose metabolism are strongly associated, as hypertriglyceridemia correlates with insulin resistance. In combination with the lower peak concentrations, it can be hypothesized that LCP-tacrolimus results in better glucose metabolism after kidney transplantation, compared to twicedaily tacrolimus Better understanding of glucose metabolism under different tacrolimus formulations would address a key component of long-term cardiovascular risk and patient outcome after kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Stable adult kidney transplant recipients on maintenance immunosuppression, >=12 months after kidney transplantation; stable is defined as no need for diagnostic and therapeutic interventions (e.g. kidney biopsy)
* Tacrolimus-based immunosuppression in combination with mycophenolic acid or azathioprine and maintenance prednisolone (<= 5 mg/q.d.) for at least 3 months
* Must be >= 18 years at the time of signing the informed consent
* Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures.
* Able to adhere to the study visit schedule and other protocol requirements.
* Subject (male or female) is willing to use highly effective methods during the study treatment (adequate: combined hormonal contraception associated with inhibition of ovulation, progestogen-only hormonal contraception associated with inhibition of ovulation, intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomized partner, sexual abstinence).
* Females of childbearing potential (FCBP) must agree to pregnancy testing within 7 days from 1st dosing of IMP
* To abstain from breastfeeding during study participation and 28 days after study drug discontinuation.
* All subjects must agree not to share medication

Exclusion Criteria:

* patients with known diabetes mellitus or PTDM, or HbA1c>=6.5%
* fasting plasma glucose on examination day (visit 1) of >= 126 mg/dl (7,0 mmol/l)
* patients with combined transplantation (e.g. liver-kidney, pancreas-kidney, etc.)
* patients with acute infection at time of baseline visit
* patients with known non-adherence
* patients with rejection therapy or increased dosis of corticosteroids for other reasons within 3 months prior to inclusion.
* Women during pregnancy and lactation.
* History of hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product.
* Participation in other interventional clinical trials (inclusive of the Follow-up period)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Difference in insulin secretion | 16 and 32 weeks
  The Difference in insulin secretion is determined by ratio AUC insulin / AUC glucose during OGTT at timepoints 16 and 32 weeks after randomization in intraindividual treatment crossover.

SECONDARY OUTCOMES:
Differences in parameters of glucose metabolism: fasting plasma glucose | 16 and 32 weeks
  Assessment of fasting plasma glucose determined in [mg/dl].
Differences in parameters of glucose metabolism: OGTT | 16 and 32 weeks
  Assessment of 2h glucose in an extended oral glucose tolerance test (OGTT) determined in [mg/dl].
Differences in parameters of glucose metabolism: insulin sensitivity | 16 and 32 weeks
  Assessment of insulin sensitivity determined in [µmol/l].
Differences in blood lipid levels | 16 and 32 weeks
  Assessment of blood lipid levels determined in [mg/dl].
Allograft function: eGFR | 16 and 32 weeks
  Assessment of eGFR (estimated glomerular filtration rate) determined in [ml/min].
Allograft function: urinary albumin excretion | 16 and 32 weeks
  Assessment of urinary albumin excretion determined in [g/dl].
Drug concentration/dose ratio | 16 and 32 weeks
  Assessment of Drug concentration/dose ratio (C/D Ratio) is determined by
  Tacrolimus level [ng/ml] related to the dose of tacrolimus taken orally the previous day [mg]:
  C/D Ratio [ng/ml x 1/mg].

CONTACTS AND LOCATIONS:
Overall Officials: Martina Guthoff, PD Dr., Principal Investigator — University Hospital Tuebingen
Locations (1):
- University Hospital Tuebingen, Tübingen, Germany